CLINICAL TRIAL: NCT06157957
Title: Lung Cancer Screening Pilot Programme: Cancer Screening Smoking Cessation AND Respiratory Assessment
Brief Title: Cancer Screening Smoking Cessation AND Respiratory Assessment
Acronym: CASSANDRA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Hospital de Sant Pau
Record Dates: First submitted 2023-11-24; First posted 2023-12-06 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer; Protection Against Malignant Lung Neoplasm (Diagnosis)
Keywords: lung cancer; tobacco cessation; respiratory assessment
MeSH Terms: conditions — Lung Neoplasms; Disease; Tobacco Use Cessation | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active smokers (Other): We do a CT scan in active smokers and ex-smokers plus an spirometry combined to a tobacco cessation programme in active smokers
  Interventions: Diagnostic Test: Lung cancer screening with low dose CT scan

INTERVENTIONS:
Diagnostic Test: Lung cancer screening with low dose CT scan — Low dose CT scan in active smokers or ex-smokers with an age between 50 and 75 years old

SUMMARY:
The CASSANDRA project (Cancer Screening, Smoking Cessation, AND Respiratory Assessment) is a project led by SEPAR whose main coordinators are Dr. Luis Seijo, a pulmonologist at the Clínica Universitaria de Navarra, and Dr. Juan Carlos Trujillo-Reyes, a thoracic surgeon at the Hospital de la Santa Creu I Sant Pau and Coordinator of the Thoracic Oncology Area, in addition to the collaboration of a large number of professionals with expertise in lung cancer screening.

Despite its proven efficacy, Spain does not yet have a unified lung cancer screening protocol. The aim of the CASSANDRA project is to initiate a national screening program that can join forces with existing smoking cessation programs in Spain, which have proven to be insufficient in reducing the number of people affected by lung cancer.

CASSANDRA aims to analyze the feasibility of implementing a lung cancer screening program in Spain implemented in the public health system and carry out a cost-effectiveness analysis

DETAILED DESCRIPTION:
CASSANDRA aims to be the first lung cancer screening pilot project in Spain. A project to assess the feasibility of implementation as well as to look for models that allow a better selection of the cases to be screened.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years active smoker with cumulative dose of >20 packets/year
* Age 50-75 years ex-smoker less than 15 years old with cumulative dose of > 20 packets/year

Exclusion Criteria:

* Pre-existing or new-onset comorbidities that, in the opinion of the coordinator, prevent surgical resection if lung cancer is found on low dose computed tomography (LDCT) scan, for example, severe chronic obstructive pulmonary disease (COPD) with forced expiratory volume at one second (FEV1) < 30%.
* Inability to sign the informed consent or collaborate with the CT scan.
* Performing a chest CT for any reason in the previous year or planned CT for any reason in the next 3 months.
* Subjects with a history of any cancer (except non-melanoma skin cancer) in the 5 years prior to inclusion in the screening program.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40000 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of lung cancer in early stage in a high risk population during a lung cancer screening programme. We measure this outcome depending on the CT results. | 0 years until 5 years
  Lung cancer screening
The number of patients who quit smoking during a lung cancer screening program. We will measure this parameter by recording smoking cessation during the 5 years. | 0 years until 5 years
  Tobacco Cessation
The number of patients who present other diseases associated with smoking such as emphysema, COPD or coronary pathology. We will measure this parameter by means of spirometry and CT scan. | 0 years until 5 years
  Respiratory assessment

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Trujillo Reyes, MD/PHD, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau

IPD SHARING:
Plan to Share IPD: Yes
We have a PI in each center enrolled to the project. More than 40 hospitals are enrolled to the CASSANDRA project
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1, 3 years after the beginning and at the end of the study
Access Criteria: PI of each centre enrolled to CASSANDRA have a passwords to access to the database
URL: http://cassandra.xolomon.com/Home?returnurl=%2f